CLINICAL TRIAL: NCT03188081
Title: A Prospective, Multicentric, Observational Study to Investigate the Effectiveness of an Education Support Program on Medication Adherence in Italian Real Life RA Patients Treated With Abatacept SC
Brief Title: A Study to Investigate the Effectiveness of an Education Support Program on Medication Adherence in Italian Real Life Rheumatoid Arthritis (RA) Patients Treated With Subcutaneous (SC) Abatacept
Acronym: TIGHT
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-645
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort A: Adult RA patients followed up according to local clinical practice only at the hospital wards
- Cohort B: Adult RA patients followed up according to local clinical practice at the Hospital wards and additionally at their home through a support program

SUMMARY:
The primary objective of this study is to investigate whether an Educational Supported Program (ESP), including tight control procedures implemented through patient home care, has positive impact in terms of better adherence to the therapy with abatacept SC at 12 months after treatment start (1st injection). In the scope of this objective the adherence is measured by the Medication Adherence Questionnaire (MAQ).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to participate in the study signed by the patient
* Age ≥ 18 years at the date of consent subscription
* Diagnosis of active Rheumatoid Arthritis moderate to severe as per the 1987 American College of Rheumatology (ACR) criteria/2010 ACR/ European League Against Rheumatism (EULAR) RA Classification Criteria
* Naïve of abatacept
* Initiated with abatacept SC either as 1st or 2nd line biologic treatment after inadequate response to previous therapy with one or more DMARDs according to Summary of Product Characteristics (SmPC) locally approved

Exclusion Criteria:

* Participating in clinical trial or other non-interventional studies, excluding registries
* Inability to read and write
* Any condition that in the investigator's opinion might jeopardize the follow-up and the data collection for the entire study observation period (24 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult RA patients, naïve of abatacept, initiated with abatacept SC either as 1st or 2nd line biologic treatment after inadequate response to previous therapy with one or more Disease-Modifying Anti-Rheumatic Drugs (DMARDs)
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Change in Medication Adherence Questionnaire (MAQ) | 12 months and 24 months
  To investigate whether an Educational Support Program (ESP), including tight control procedures implemented through patient home care, has positive impact in terms of better adherence to the therapy with abatacept SC at 12 months and 24 months after treatment start (1st injection)
Adherence ratio | 24 months
  Percentage ratio between the total number of injections taken in a treatment period and the total number of injections expected to be taken in the same treatment period according to rheumatologist prescription

SECONDARY OUTCOMES:
Distribution of socio-demographic data | 24 months
  To describe the major characteristics of population of patients in real life conditions at abatacept SC initiation
Patient Rheumatoid Arthritis History | 24 months
  To describe the major characteristics of population of patients in real life conditions at abatacept SC initiation
Co-morbidities | 24 months
  To describe the major characteristics of population of patients in real life conditions at abatacept SC initiation
Clinical measurements (disease indices and relevant subcomponents) | 24 months
  To describe the major characteristics of population of patients in real life conditions at abatacept SC initiation
Erythrocyte Sedimentation Rate | 24 months
  To describe the major characteristics of population of patients in real life conditions at abatacept SC initiation
Rheumatoid Factor | 24 months
  To describe the major characteristics of population of patients in real life conditions at abatacept SC initiation
Anti Citrullinated Peptide Antibody | 24 months
  To describe the major characteristics of population of patients in real life conditions at abatacept SC initiation
Prior RA treatments | 24 months
  To describe the major characteristics of population of patients in real life conditions at abatacept SC initiation
Patient's reported assessment of health measured by HAQ-DI | 24 months
  To describe the major characteristics of population of patients in real life conditions at abatacept SC initiation and to investigate whether a better adherence to the abatacept SC therapy is associated to a better health status of the patient population
Health related quality of life measured by EQ-5D | 24 months
  To describe the major characteristics of population of patients in real life conditions at abatacept SC initiation and to investigate whether a better adherence to the abatacept SC therapy is associated to a better health status of the patient population
Remission rate measured by MAQ | 24 months
  To investigate whether a better adherence to the abatacept SC therapy is associated to a better clinical outcome of the patient population
Low disease activity rate measured by MAQ | 24 months
  To investigate whether a better adherence to the abatacept SC therapy is associated to a better clinical outcome of the patient population
DAS28 score measured by MAQ | 24 months
  To investigate whether a better adherence to the abatacept SC therapy is associated to a better clinical outcome of the patient population
Concomitant medication for RA (Synthetic DMARDs and corticosteroids) | 24 months
  To describe the use of concomitant medication for RA (Synthetic DMARDs and corticosteroids) over the study observation period
Adverse Events | 24 months
  To describe the incidence of Adverse Events, by seriousness and relationship with abatacept SC
Reason for Withdrawal, where applicable | 24 months
  To describe the incidence of the reasons for withdrawal from the treatment and the study
Retention rate | 24 months
  To evaluate the retention rate calculated as the time-to-discontinuation of abatacept SC treatment over the study observation period
Cost-utility analysis (CUA) | 24 months
  To perform a cost-utility analysis (CUA) from the National Health System
Societal perspective comparing health consequences | 24 months
  Societal perspective comparing health consequences Quality Adjusted Life Years (QALYs)
Cost of alternative follow-up strategies | 24 months
  Two alternative follow-up strategies: ESP versus standard control
Patient's reported assessment of health measured by Pain VAS | 24 months
  To describe the major characteristics of population of patients in real life conditions at abatacept SC initiation and to investigate whether a better adherence to the abatacept SC therapy is associated to a better health status of the patient population

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Brescia, Italy

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm